CLINICAL TRIAL: NCT03609723
Title: Combined Use of a Novel Cardioplegic Formula With MPS ® Using the MiECC in Isolated CABG Versus OPCABG
Acronym: OPCBAG
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00923; ch18reuthebuch2
Record Dates: First submitted 2018-07-17; First posted 2018-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Complication of Coronary Artery Bypass Graft; Complication of Extracorporeal Circulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MPS® in patients with CABG: Patients undergoing coronary artery bypass grafting with application of a myocardial protection system (MPS ®) and using a minimal extracorporeal circulation system (MiECC)
  Interventions: Procedure: CABG
- OPCABG in patients with CABG: Patients undergoing coronary artery bypass grafting without use of a minimal extracorporeal circulation system (Off-pump coronary artery bypass grafting = OPCABG)
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: CABG — CABG with application of a myocardial protection system (MPS ®) and using a minimal extracorporeal circulation system (MiECC) or CABG without use of a minimal extracorporeal circulation system (Off-pump coronary artery bypass grafting = OPCABG)

SUMMARY:
A patient group receiving a novel cardioplegic formula with MPS ® (Myocardial protection system) and using the MiECC (Minimal extracorporeal circulation system) when undergoing coronary artery bypass grafting is compared to a retrospective patient group undergoing Off-pump coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* CABG using MPS® or OPCABG

Exclusion Criteria:

* use of other colloid solution than Cardioplexol ® for MPS®
* other inventions than CABG
* myocardial infarction <7 days before CABG
* patients denial of data use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing coronary artery bypass grafting with application of a myocardial protection system (MPS ®) and using a minimal extracorporeal circulation system (MiECC) Patients undergoing coronary artery bypass grafting without use of a minimal extracorporeal circulation system (Off-pump coronary artery bypass grafting = OPCABG)
Sampling Method: Probability Sample
Enrollment: 2433 (Actual)
Dates: Start 2010-06-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
assessment of cardial biomarkers as high sensitive troponin T (hs-TrT), Creatinkinase (CK) and Creatinkinase myocardial type (CK-MB) | perioperative during hospital stay for CABG
  high sensitive troponin T (hs-TrT), Creatinkinase, (CK) Creatinkinase myocardial type (CK-MB)

SECONDARY OUTCOMES:
mortality | 30 days after CABG
  death after coronary artery bypass grafting
need for intensive care unit | perioperative during hospital stay for CABG
  duration of stay at intensive care unit
occurence of dysrhythmia | perioperative during hospital stay for CABG
  rhythm disturbance after CABG

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Reuthebuch, PD MD, Principal Investigator — Klinik für Herzchirurgie, Universitätsspital Basel Spitalstrasse 21 4031 Basel
Locations (1):
- Herzchirurgie University Hospital Basel, Basel, Switzerland